CLINICAL TRIAL: NCT01988467
Title: The Protective Role of the Nose During Acute Exposure to Passive Smoking.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hellenic Anticancer Society (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6322/6.3.13
Record Dates: First submitted 2013-10-28; First posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Second Hand Smoke Exposure
Keywords: nasal breathing, oral breathing, secondhand smoking,

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nasal breathing (Experimental): At the time that the exposure took place with nasal breathing, the study was as follows:
  Before the exposure: rhinomanometry, IOS , FeNO , spirometry, plethysmography, P.100.
  Exposure to second hand smoking:Each volunteer was exposed to secondhand smoking twice, for 20 minutes, once with nasal breathing and once with oral breathing, with 3 days interval and in random sequence.
  After the exposure: rhinomanometry, IOS , FeNO , spirometry,plethysmography , P.100.
  Interventions: Other: exposure to second hand smoking
- oral breathing (Experimental): At the time that the exposure took place with oral breathing, the study was as follows:
  Before the exposure: IOS, exhaled nitric oxide (FeNO), spirometry, plethysmography and P.100.
  Exposure to second hand smoking: each volunteer was exposed to secondhand smoking twice, for 20 minutes, once with nasal breathing and once with oral breathing, with 3 days interval and in random sequence.
  After the exposure: IOS, FeNO, spirometry,plethysmography and P.100.
  Interventions: Other: exposure to second hand smoking

INTERVENTIONS:
Other: exposure to second hand smoking — The duration of the exposure to second hand smoke both days was for 20 minutes within a 250mgr/m3 concentration box room. A smoking machine was used, which mimics the smoker (up to 6 breaths per minute in tobacco volume 80ml for each inhalation). The exposure was sometimes with closed mouth and others with closed nose in random sequence.

SUMMARY:
The aim of this study was to compare the acute effects of second hand smoke exposure between nasal and oral breathing and to assess the potential protective role of the nose during acute exposure, in exposure conditions similar to those within a bar where smoking is permitted.

DETAILED DESCRIPTION:
Analysis of the laboratory testing:

The measurement of NO for the respiratory tract was performed with a Ecomedics CLD 88spNO analyzer as follows: the examinee performed tidal breathing with a closed nose, through a special mouthpiece and then took a deep breath and exhale steadily with a flow of 50ml/sec. After 3 attempts, during which we obtained an exhaled NO measurement each time, until we obtained a reliability index CV <10%.

For the oscillometry (IOS) of the respiratory tract the Master Screen IOS VIASYS was used, the examinee breathed quietly through the mouthpiece with his/her nose closed for a period of 1 minute. In this way we measured the impedance Z at 5 Hz, the resistance to 5,10,20 Hz respectively, the reactance in 5,10,20 Hz respectively, the central and peripheral airway resistance and resonant frequency.

Rhinomanometry was done by the Master Screen IOS VIASYS system, the examinee breathed calmly through the examined nostril, while the other was closed, 5 breaths per attempt were performed. After 3 attempts for each nostril, we assessed the average inspiratory resistance for each nostril separately.

The plethysmography took place on the Master Screen Body of VIASYS, the door of the Body was closed as well as all the doors of the room and without the presence of motion in the test room. The subject performed calm breaths with a closed nose, through the mouthpiece and then took a deep breath, followed by deep exhalation. At the end of the effort we had values for the total lung capacity (TLC), residual volume (RV), airway resistance (R), vital capacity (VC), the functional residual capacity (FRC), Exhaled residual volume (ERV) and the ratio RV / TLC. This was repeated 3 times and one was selected to be the most representative.

The P.100 was performed through the Master Screen Body of VIASYS with the door of the Body Box opened. The volunteer was performing calm breaths with a closed nose, through the mouthpiece, during which a shutter blocked the flow. The obtained value of the pressure was the one that developed in the first second of inhalation with the shutter down is noted. This repeated 3 times and one selected to be the most representative.

Spirometry and the flow-volume curve were assessed with a Master Screen Body of VIASYS with the door of the Body Box opened as follows: The subject performed tidal breathing with a closed nose, through the mouthpiece, and then took a sharp deep breath, which was followed by sharp deep exhalation, and the test ended with deep inhalation. At the end of the effort we had values for forced vital capacity (FVC), the violent expiratory the first volume 1 (FEV1), the ratio FVC/FEV1%, peak expiratory flow (PEF) and mesoexpiratory flow in peripheral airways than 25% to 75% of vital capacity. This was repeated 3 times and one was selected to be the most representative.

The assessment of the type of breathing during exposure to secondhand smoke was performed through the VIASYS Respitrace. The protocol was as follows: The volunteer breathed calmly over 20 times with the mouth closed and once with a closed nose, while wearing two rubber bands, one on the chest and one to the abdomen, which incorporates electrodes. The waveform of the breath in the thorax, abdomen and the average of these was recorded in real time. Also, for every breath we had values for the inspiratory time, expiratory time, total time, the participation rate of the chest, the participation rate of the ventricle, the peak inspiratory flow (Pif), the mean inspiratory flow (Mif), and the flow-volume curve and the analysis chart of each breath in the thoracic and abdominal component.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer adults non-smokers

Exclusion Criteria:

* < 18 years old
* Recent or chronic disease of the upper or lower respiratory system.
* Current pregnancy
* Breastfeeding women

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
exhaled nitric oxide (FeNO) for the respiratory tract | before exposure (Baseline) and after exposure with a 30 minutes interval
  To compare the changes between the two types of breathing
plethysmography | before exposure (Baseline) and after exposure with a 30 minutes interval
  plethysmography take place both at oral and nasal breathing twice before and after intervention.

SECONDARY OUTCOMES:
Eye or nose irritation | during the exposure to second hand smoke
  During the exposure to second hand smoke that lasted 20 minutes the examinee had his /her mouth closed and filled in an evaluation Questionnaire about eye or nose irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis K Behrakis, Professor, Study Chair — National and Kapodistrian University of Athens; Palagia M Karas, MD, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- Hellenic Anticancer Society, Athens, Attica, Greece

REFERENCES:
- [Background] Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Acute pulmonary effects of sidestream secondhand smoke at simulated car concentrations. Xenobiotica. 2013 Jun;43(6):509-13. doi: 10.3109/00498254.2012.741272. Epub 2012 Dec 4. PMID 23205567
- [Background] Vardavas CI, Anagnostopoulos N, Kougias M, Evangelopoulou V, Connolly GN, Behrakis PK. Short-term pulmonary effects of using an electronic cigarette: impact on respiratory flow resistance, impedance, and exhaled nitric oxide. Chest. 2012 Jun;141(6):1400-1406. doi: 10.1378/chest.11-2443. Epub 2011 Dec 22. PMID 22194587